CLINICAL TRIAL: NCT05005754
Title: An Interventional Study for the Beneficial Effects of Probiotics on Cardio-metabolic Health in Chinese Subjects
Brief Title: Effect of Probiotics on Cardiometabolic Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Min Xia, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Pro-2021
Record Dates: First submitted 2021-08-08; First posted 2021-08-16 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Cardiometabolic Risk Factors
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics (Experimental): Subjects are instructed to take one capsule of probiotics daily for a total of 3 months
  Interventions: Dietary Supplement: Probiotics
- Placebo Control (Placebo Comparator): Subjects are instructed to take one capsule of placebo daily for a total of 3 months
  Interventions: Dietary Supplement: Placebo control

INTERVENTIONS:
Dietary Supplement: Probiotics — During the study period, subjects are instructed to take one capsule of probiotics daily for a total of 3 months. Aside from the probiotic supplement, all participants are instructed to continue their normal routine and not make any changes to their habitual diet or exercise habits.
  Arms: Probiotics
Dietary Supplement: Placebo control — During the study period, subjects are instructed to take one capsule of placebo control daily for a total of 3 months. Aside from the probiotic supplement, all participants are instructed to continue their normal routine and not make any changes to their habitual diet or exercise habits.
  Arms: Placebo Control

SUMMARY:
Atherosclerosis is a major risk factor for cardiovascular diseases. Recently, dysbiosis of gut microbiota has been reported to play an important role in the pathogenesis of atherosclerosis. Animal studies have demonstrated that administration of probiotics help delay the progression of atherosclerosis through several mechanisms. This trial aims to examine its protective effect in humans.

DETAILED DESCRIPTION:
Atherosclerosis is a major risk factor for cardiovascular diseases. Recently, dysbiosis of gut microbiota has been reported to play an important role in the pathogenesis of atherosclerosis. Animal studies have demonstrated that administration of probiotics help delay the progression of atherosclerosis through several mechanisms such as reduction in endotoxemia, and enhanced production of short-chain fatty acids.

However, whether administration of probiotics also has a protective effect in subjects with metabolic syndrome (MetS), who are at high risk for developing atherosclerosis, remain unknown.

ELIGIBILITY:
Inclusion Criteria:

* Local residents aged between 30-60 years old;
* Stable weight (<5% weight change over last 3 months);
* Central obesity defined as waist circumference ≥90 cm in males or ≥80 cm in females, Plus any two of the following four conditions i) Elevated triglycerides: serum triglycerides ≥150 mg/dL (1.7 mmol/L); ii) Reduced HDL cholesterol: serum HDL-c <40 mg/dL (1.03 mmol/L) in males or <50 mg/dL (1.29 mmol/L) in females; iii) Elevated blood pressure: systolic blood pressure ≥130 mmHg or diastolic blood pressure ≥85 mmHg; iv) Elevated fasting plasma glucose: fasting plasma glucose ≥100 mg/dL (5.6 mmol/L)
* Absence of any systemic, cardiovascular diseases, as well as infections within the previous month;
* Absence of any diet or medication that might interfere with metabolic homoeostasis and gut microbiota, especially antibiotics and probiotics 4 weeks before recruitment.

Exclusion Criteria:

* Acute illness or current evidence of acute or chronic inflammatory of infective diseases;
* Participation in regular diet program more than 2 times per week in the latest 3 months prior to recruitment;
* Mental illness rendering them unable to understand the nature, scope, and possible consequences of the study.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Flow-mediated slowing (FMS) | from baseline to 12 weeks after intervention
  FMS is a simple test for endothelial functions measured by Vicorder. In patients whose endothelial function or flow-mediated vasodilation are compromised, the FMS is substantially reduced.

SECONDARY OUTCOMES:
gut microbiota | from baseline to 12 weeks after intervention
  Alterations of the composition of gut microbiota evaluated by metagenomics
microbial metabolites | from baseline to 12 weeks after intervention
  alterations of microbial metabolites evaluated by High performance liquid chromatography-mass spectrometry
Metabolic Syndrome Severity Z Score (MetZ score) | from baseline to 12 weeks after intervention
  MetZ score is an weighted score of the five traditional components of Metabolic syndrome (waist, triglyceride, HDL cholesterol, SBP and fasting glucose). It's used to evaluate the severity of metabolic disorder, and a higher score indicates a more severe status.
Lipid profiles | from baseline to 12 weeks after intervention
  alterations of blood lipids including total cholesterol, triglyceride, LDL cholesterol and HDL cholesterol determined by automatic biochemical analyser
Blood pressure | from baseline to 12 weeks after intervention
  alterations of blood pressure
Insulin sensitivity | from baseline to 12 weeks after intervention
  alterations of HOMA-IR index

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Department of Nutrition and Food Hygiene, Guangzhou, Guangdong
  - Sun Yat-Sen University, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang J, Huang J, Huang Z, Xu Y, Li W, Zhu S, Zhao Y, Ye B, Liu L, Zhu J, Xia M, Liu Y. Cardiometabolic benefits of Lacticaseibacillus paracasei 8700:2: A randomized double-blind placebo-controlled trial. Clin Nutr. 2023 Sep;42(9):1637-1646. doi: 10.1016/j.clnu.2023.07.017. Epub 2023 Jul 21. PMID 37506599